CLINICAL TRIAL: NCT01512095
Title: A Trial to Examine the Bioequivalence of Norditropin® Versus Nutropin AQ® in Healthy Adult Volunteers
Brief Title: Bioequivalence of Two Products (Norditropin® Versus Nutropin AQ®) in Healthy Adult Volunteers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GH-3958; 2012-003381-40 (EudraCT Number); U1111-1122-9661 (Other: WHO)
Record Dates: First submitted 2012-01-09; First posted 2012-01-19 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2013-09

CONDITIONS: Growth Disorder; Healthy
MeSH Terms: conditions — Growth Disorders | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Norditropin® (Experimental)
  Interventions: Drug: somatropin
- Nutropin AQ® (Active Comparator)
  Interventions: Drug: somatropin

INTERVENTIONS:
Drug: somatropin — A single dose administered subcutaneously (under the skin) on 2 separate dosing visits (treatment periods) separated by a wash-out period
  Arms: Norditropin®
Drug: somatropin — A single dose administered subcutaneously (under the skin) on 2 separate dosing visits (treatment periods) separated by a wash-out period
  Arms: Nutropin AQ®

SUMMARY:
This trial is conducted in Europe and United States of America (USA). The aim of this trial is to examine the bioequivalence (assessment of the expected biological equivalence of two pharmaceutical drug products with identical active ingredient) of Norditropin® versus Nutropin AQ® in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* No previous exposure to recombinant human GH (growth hormone)or IGF-I (insulin-like growth factor-I)
* Body mass index (BMI) 18.0-27.0 kg/m^2 (both inclusive)
* Considered generally healthy upon completion of medical history, physical examination, vital signs, screening laboratory results, and electrocardiogram (ECG), as judged by the Investigator

Exclusion Criteria:

* The receipt of any investigational medicinal product within 1 month prior to this trial
* Current or previous treatment with recombinant human growth hormone or IGF-I
* Female of childbearing potential who is pregnant, breast-feeding or intends to become pregnant or is not using adequate contraceptive methods (adequate contraceptive measures as required by local law) for the duration of the trial
* Known presence or history of malignancy
* Diabetes mellitus
* Use of pharmacologic doses of glucocorticoids
* Use of anabolic steroids
* History of drug or alcohol abuse

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2013-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Area under the serum hGH (human growth hormone) concentration-time curve (AUC0-t) | From 0 to the time of the last quantifiable concentration over a 24-hour sampling period
Maximum observed serum hGH concentration | Over a 24-hour sampling period
Area under the effect (IGF-I) curve from time 0 to the time of the last concentration (AUEC0-t) | Over a 96-hour sampling period
Maximum IGF-I (insulin-like growth factor-I) effect (Emax) | Over a 96-hour sampling period

SECONDARY OUTCOMES:
The frequency of adverse events (AE) and vital signs | From screening (14 days before randomisation) to follow-up period (3-21 days after randomisation)
The frequency of abnormal hematology | From screening (14 days before randomisation) to follow-up period (20-23 days after randomisation)
The frequency of abnormal findings in physical examinations | From screening (14 days before randomisation) to follow-up period (20-23 days after randomisation)
Biochemistry laboratory parameters | From screening (14 days before randomisation) to follow-up period (20-23 days after randomisation)
The frequency of injection site reaction | From the time of injection of the trial product (day 1 and day 13) to follow-up during the two dosing periods (day 5 and day 17)
Area under the effect (IGFBP-3) curve | From time 0 to the time of the last concentration (AUEC0-t) over a 96-hour sampling period
Maximum IGFBP-3 (insulin-like growth factor binding protein 3) effect (Emax) | Over a 96-hour sampling period

CONTACTS AND LOCATIONS:
Overall Officials: John Germak, Study Director — Novo Nordisk A/S

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com